CLINICAL TRIAL: NCT02428647
Title: Lao Zinc Study: The Effects of Two Forms of Daily Preventive Zinc Supplementation Versus Therapeutic Zinc Supplementation for Diarrhea on Young Children's Physical Growth and Risk of New Episodes of Diarrhea
Brief Title: Lao Zinc Study: Effects of Two Forms of Daily Preventive Zinc Versus Therapeutic Zinc Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Lao Tropical and Public Health Institute, Lao PDR (Unknown); USDA, Western Human Nutrition Research Center (U.S. Federal Agency); University of British Columbia (Other); Khon Kaen University (Other); Nutrition International (Other); The Mathile Institute for the Advancement of Human Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 626187; 10-1347-UCALIF-07 (Other: Other)
Record Dates: First submitted 2015-02-09; First posted 2015-04-29 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Diarrhea
Keywords: growth; plasma zinc concentration
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- micronutrient powder (MNP) (Active Comparator): preventive zinc supplements provided as MNP (containing 10 mg zinc and 14 other nutrients, including 6 mg iron, 0.56 mg copper, 17 μg selenium, 90 μg iodine, 400 μg RE vitamin A, 5 μg vitamin D, 5 mg vitamin E, 30 mg ascorbic acid, 0.5 mg vitamin B1, 0.5 mg vitamin B2, 6 mg niacin, 0.5 mg vitamin B6, 0.9 μg vitamin B12, and 150 μg folate,) plus ORS and therapeutic placebo supplements for diarrhea
  Interventions: Dietary Supplement: MNP; Dietary Supplement: therapeutic placebo supplement
- placebo powder (Placebo Comparator): placebo powder plus ORS and therapeutic placebo supplements for diarrhea
  Interventions: Dietary Supplement: therapeutic placebo supplement; Dietary Supplement: placebo powder
- preventive zinc supplements (Active Comparator): preventive zinc supplements provided as dispersible zinc tablets (containing 7 mg zinc, to be given between meals) plus ORS and therapeutic placebo supplements for diarrhea
  Interventions: Dietary Supplement: preventive zinc supplement; Dietary Supplement: therapeutic placebo supplement
- therapeutic zinc supplements (Active Comparator): preventive placebo supplements provided as dispersible tablets plus ORS and dispersible therapeutic zinc tablets (containing 20 mg zinc) for diarrhea
  Interventions: Dietary Supplement: therapeutic zinc supplement; Dietary Supplement: preventive placebo supplement

INTERVENTIONS:
Dietary Supplement: MNP — MNP containing containing 10 mg zinc and 14 other nutrients, including 6 mg iron, 0.56 mg copper, 17 μg selenium, 90 μg iodine, 400 μg RE vitamin A, 5 μg vitamin D, 5 mg vitamin E, 30 mg ascorbic acid, 0.5 mg vitamin B1, 0.5 mg vitamin B2, 6 mg niacin, 0.5 mg vitamin B6, 0.9 μg vitamin B12, and 150 μg folate
  Arms: micronutrient powder (MNP)
Dietary Supplement: preventive zinc supplement — 7 mg zinc daily as dispersible tablet
  Arms: preventive zinc supplements
Dietary Supplement: therapeutic zinc supplement — 20 mg zinc per day for 10 days during diarrhea episodes, as dispersible tablet
  Arms: therapeutic zinc supplements
Dietary Supplement: preventive placebo supplement — dispersible daily placebo tablet
  Arms: therapeutic zinc supplements
Dietary Supplement: therapeutic placebo supplement — dispersible placebo tablet for 10 days during diarrhea episodes
  Arms: micronutrient powder (MNP); placebo powder; preventive zinc supplements
Dietary Supplement: placebo powder — placebo powder
  Arms: placebo powder

SUMMARY:
The study will be conducted as a community-based, randomized, placebo-controlled, trial with four study groups. The overall objective of the study is to determine the optimal method for delivering zinc to young children, both for the prevention of zinc deficiency and treatment of diarrhea. In particular, the investigators plan to compare the impact on physical growth, morbidity, micronutrient status, immune function, environmental enteric dysfunction, parasite burden and hair cortisol concentration of: 1) daily preventive zinc supplementation as a micronutrient powder (MNP); 2) placebo powders; 3) daily preventive zinc supplementation as dispersible tablets; 4) therapeutic zinc supplementation as dispersible tablets given in relation to episodes of diarrhea.

In addition to the major outcomes mentioned above, the investigators will monitor adherence to the interventions, neuro-behavioral development, and the occurrence of any adverse events.

DETAILED DESCRIPTION:
Zinc is an essential nutrient that is required for children's normal growth and resistance to infections, including diarrhea and pneumonia, two major causes of child mortality. Current strategies for controlling the growth and infection-related complications of zinc deficiency include: 1) daily or weekly preventive zinc supplementation, and 2) therapeutic zinc supplementation for 10-14 days in relation to episodes of diarrhea. Information is needed on the relative impact of these intervention strategies on children's growth and risk of new episodes of diarrhea (and other infections).

Preventive zinc supplements can be delivered either as a single nutrient (zinc) supplement or as a multiple micronutrient (MMN) supplement, such as micronutrient powders (MNP) added to young children's complementary food. Available research indicates that zinc delivered in MNP at the currently recommended dose (4.1-5 mg/d) has not had a measurable impact on zinc-related functional outcomes, like growth and prevention of infection. Moreover, some studies of MMN supplements have detected a greater incidence of diarrhea in the MMN group than in the non-intervention or placebo control groups. Thus, despite the beneficial effects of MNP on prevention of anemia and enhancing iron status, questions have been raised about the desirability of providing zinc in MNP (containing iron and other nutrients) versus a single nutrient formulation offered between meals. For these reasons, the present study is designed to compare both the zinc delivery plan (i.e., preventive versus therapeutic supplementation) as well as the form of delivering zinc (i.e., as a dispersible tablet given between meals or as a MNP given with meals) and to permit assessment of any adverse effects of MNP on the incidence of diarrhea.

The study will be conducted as a community-based, randomized, placebo-controlled trial with four study groups in rural communities of Khammouane Province in Central Lao PDR.

The project team will enroll a total of ~3,400 children whose ages will range from 6-23 months. Children will be randomly assigned to one of four study group: 1) preventive zinc supplementation provided as LI-MNP plus ORS and placebo tablets for treatment of diarrhea; 2) placebo preventive supplementation provided as placebo powder plus ORS and placebo tablets for diarrhea ; 3) preventive zinc supplementation provided as dispersible zinc tablets (containing 7 mg zinc, to be given between meals) plus ORS and placebo tablets for diarrhea; and 4) therapeutic zinc supplementation provided as dispersible tablets (containing 20 mg zinc) for diarrhea plus ORS and placebo preventive tablets.

The major outcomes that will be monitored include adherence to the interventions; physical growth; incidence, duration and severity of episodes of diarrhea; changes in MN status; immune function; environmental enteric dysfunction; parasite burden; hair cortisol concentration; neuro-behavioral development; and the occurrence of any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from at least one parent or primary caregiver
* Age 6-23 months initially
* Permanent resident of study area
* Planned availability during the period of the study
* Acceptance of home visitors

Exclusion Criteria:

* Weight-for-height z-score (WHZ) <-3Z with respect to WHO 2006 standards
* Presence of bipedal edema
* Severe illness warranting hospital referral
* Congenital abnormalities potentially interfering with growth
* Chronic medical condition (e.g. malignancy) requiring frequent medical attention
* Known HIV infection of index child or child's mother
* Hemoglobin <70 g/L
* Currently consuming zinc supplements
* Current participation in any other clinical trial

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3433 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in length and length-for-age Z-score | 36 weeks
Change in weight and weight-for-age Z-score | 36 weeks
Incidence of diarrhea | 36 weeks
Change in hemoglobin concentration | 32 weeks
Change in micronutrient status | 32 weeks
  plasma zinc, ferritin, transferrin receptor; and retinol binding protein (RBP) concentrations, measured in a subsample of 560 participants, and controlling for the presence of elevated acute phase protein
Innate and adaptive immune defense | 32 weeks
  production of cytokines by cultures of peripheral blood white blood cells; and change in concentrations of naïve and memory CD4 and CD8 T-cells and regulatory (Treg) T-cells in a sub-set of 500 children

SECONDARY OUTCOMES:
Change in mid-upper circumference | 36 weeks
Achievement of gross motor developmental milestones | after 4, 8, 12, 16, 20, 24, 32 and 36 weeks
  Gross motor developmental milestones as recommended by the World Health Organization include: sitting without support, crawling, standing with assistance, walking with assistance, standing alone, walking alone
Change in stool calprotectin concentration | 36 weeks
Change in stool neopterin concentration | 36 weeks
Change in hair cortisol concentration | 36 weeks
Intestinal protozoa parasite infection | 36 weeks
  Intestinal protozoan infections will be assessed by a modified formalin-ethyl acetate concentration technique
Helminths parasite infection | 36 weeks
  Helminth parasite infections will be assessed using duplicate Kato-Katz thick smears
Acute and chronic sleep pattern | after 4, 8, 12, 16, 20, 24, 32 and 36 weeks
  Assessed by Brief Infant Child Sleep Questionnaire
B-vitamin status | 36 weeks
  erythrocyte thiamine diphosphate, plasma folate and B12 concentrations and erythrocyte glutathione reductase activation coefficient (EGRac) measured in a randomly selected sub-sample of 260 children (MNP and control group only)

OTHER OUTCOMES:
Incidence of serious adverse events | 36 weeks
  Serious adverse events, including death and required overnight stay in a health facility
Incidence of any non-serious adverse events | 36 weeks
  non-serious adverse events that may be detected retrospectively, such as the incidence of diarrhea, vomiting, etc., based on the results of morbidity surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Y Hess, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Lao Tropical and Public Health Institute, Vientiane, Laos

IPD SHARING:
Plan to Share IPD: Yes
The complete de-identified dataset will be made publicly available within 3 years after completion of data collection. Associated data dictionaries will be made available along with the datasets.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Summer 2020
Access Criteria: Publicly available
URL: https://osf.io/5bq9c/

REFERENCES:
- [Background] Wessells KR, Brown KH, Kounnavong S, Barffour MA, Hinnouho GM, Sayasone S, Stephensen CB, Ratsavong K, Larson CP, Arnold CD, Harding KB, Reinhart GA, Lertmemongkolchai G, Fucharoen S, Bernstein RM, Hess SY. Comparison of two forms of daily preventive zinc supplementation versus therapeutic zinc supplementation for diarrhea on young children's physical growth and risk of infection: study design and rationale for a randomized controlled trial. BMC Nutr. 2018 Nov 29;4:39. doi: 10.1186/s40795-018-0247-6. eCollection 2018. PMID 32153900
- [Result] Hess SY, Hinnouho GM, Barffour MA, Bounheuang B, Arnold CD, Bell D, Marts TH, Kounnavong S. First Field Test of an Innovative, Wider Tape to Measure Mid-Upper Arm Circumference in Young Laotian Children. Food Nutr Bull. 2018 Mar;39(1):28-38. doi: 10.1177/0379572117742502. Epub 2017 Dec 19. PMID 29258337
- [Result] Hinnouho GM, Barffour MA, Wessells KR, Brown KH, Kounnavong S, Chanhthavong B, Ratsavong K, Kewcharoenwong C, Hess SY. Comparison of haemoglobin assessments by HemoCue and two automated haematology analysers in young Laotian children. J Clin Pathol. 2018 Jun;71(6):532-538. doi: 10.1136/jclinpath-2017-204786. Epub 2017 Dec 2. PMID 29197856
- [Result] Kingchaiyaphum B, Sanchaisuriya K, Fucharoen G, Chaibunruang A, Hess SY, Hinnouho GM, Barffour MA, Wessells KR, Kounnavong S, Fucharoen S. Hemoglobins F, A2 , and E levels in Laotian children aged 6-23 months with Hb E disorders: Effect of age, sex, and thalassemia types. Int J Lab Hematol. 2020 Jun;42(3):277-283. doi: 10.1111/ijlh.13164. Epub 2020 Feb 12. PMID 32048804
- [Result] Wessells KR, Hinnouho GM, Barffour MA, Arnold CD, Kounnavong S, Kewcharoenwong C, Lertmemongkolchai G, Schuster GU, Stephensen CB, Hess SY. Impact of Daily Preventive Zinc or Therapeutic Zinc Supplementation for Diarrhea on Plasma Biomarkers of Environmental Enteric Dysfunction among Rural Laotian Children: A Randomized Controlled Trial. Am J Trop Med Hyg. 2020 Feb;102(2):415-426. doi: 10.4269/ajtmh.19-0584. PMID 31889508
- [Result] Hess SY, Wessells KR, Hinnouho GM, Barffour MA, Sanchaisuriya K, Arnold CD, Brown KH, Larson CP, Fucharoen S, Kounnavong S. Iron status and inherited haemoglobin disorders modify the effects of micronutrient powders on linear growth and morbidity among young Lao children in a double-blind randomised trial. Br J Nutr. 2019 Oct 28;122(8):895-909. doi: 10.1017/S0007114519001715. PMID 31303184
- [Result] Hinnouho GM, Bernstein RM, Barffour MA, Arnold CD, Wessells KR, Ratsavong K, Bounheuang B, Kounnavong S, Hess SY. Impact of Two Forms of Daily Preventive Zinc or Therapeutic Zinc Supplementation for Diarrhea on Hair Cortisol Concentrations Among Rural Laotian Children: A Randomized Controlled Trial. Nutrients. 2018 Dec 27;11(1):47. doi: 10.3390/nu11010047. PMID 30591656
- [Result] Barffour MA, Hinnouho GM, Kounnavong S, Wessells KR, Ratsavong K, Bounheuang B, Chanhthavong B, Sitthideth D, Sengnam K, Arnold CD, Brown KH, Hess SY. Effects of Daily Zinc, Daily Multiple Micronutrient Powder, or Therapeutic Zinc Supplementation for Diarrhea Prevention on Physical Growth, Anemia, and Micronutrient Status in Rural Laotian Children: A Randomized Controlled Trial. J Pediatr. 2019 Apr;207:80-89.e2. doi: 10.1016/j.jpeds.2018.11.022. Epub 2018 Dec 21. PMID 30580974
- [Result] Wessells KR, Brown KH, Arnold CD, Barffour MA, Hinnouho GM, Killilea DW, Kounnavong S, Hess SY. Plasma and Nail Zinc Concentrations, But Not Hair Zinc, Respond Positively to Two Different Forms of Preventive Zinc Supplementation in Young Laotian Children: a Randomized Controlled Trial. Biol Trace Elem Res. 2021 Feb;199(2):442-452. doi: 10.1007/s12011-020-02163-2. Epub 2020 Apr 30. PMID 32356207
- [Result] Hinnouho GM, Wessells KR, Barffour MA, Sayasone S, Arnold CD, Kounnavong S, Hess SY. Impact of Different Strategies for Delivering Supplemental Zinc on Selected Fecal Markers of Environmental Enteric Dysfunction among Young Laotian Children: A Randomized Controlled Trial. Am J Trop Med Hyg. 2020 Oct;103(4):1416-1426. doi: 10.4269/ajtmh.20-0106. PMID 32618258
- [Result] Barffour MA, Hinnouho GM, Wessells KR, Kounnavong S, Ratsavong K, Sitthideth D, Bounheuang B, Sengnam K, Chanhthavong B, Arnold CD, Brown KH, Larson CP, Hess SY. Effects of therapeutic zinc supplementation for diarrhea and two preventive zinc supplementation regimens on the incidence and duration of diarrhea and acute respiratory tract infections in rural Laotian children: A randomized controlled trial. J Glob Health. 2020 Jun;10(1):010424. doi: 10.7189/jogh.10.010424. PMID 32612816
- [Result] Kewcharoenwong C, Schuster GU, Wessells KR, Hinnouho GM, Barffour MA, Kounnavong S, Brown KH, Hess SY, Samer W, Tussakhon I, Peerson JM, Lertmemongkolchai G, Stephensen CB. Daily Preventive Zinc Supplementation Decreases Lymphocyte and Eosinophil Concentrations in Rural Laotian Children from Communities with a High Prevalence of Zinc Deficiency: Results of a Randomized Controlled Trial. J Nutr. 2020 Aug 1;150(8):2204-2213. doi: 10.1093/jn/nxaa037. PMID 32119742
- [Derived] Kewcharoenwong C, Sein MM, Nithichanon A, Khongmee A, Wessells KR, Hinnouho GM, Barffour MA, Kounnavong S, Hess SY, Stephensen CB, Lertmemongkolchai G. Daily preventive zinc supplementation increases the antibody response against pathogenic Escherichia coli in children with zinc insufficiency: a randomised controlled trial. Sci Rep. 2022 Sep 27;12(1):16084. doi: 10.1038/s41598-022-20445-8. PMID 36167891
- [Derived] Hinnouho GM, Hampel D, Shahab-Ferdows S, Barffour MA, McAnena L, Arnold CD, Ryan Wessells K, Kounnavong S, Allen LH, McNulty H, Hess SY. Daily supplementation of a multiple micronutrient powder improves folate but not thiamine, riboflavin, or vitamin B12 status among young Laotian children: a randomized controlled trial. Eur J Nutr. 2022 Oct;61(7):3423-3435. doi: 10.1007/s00394-022-02890-3. Epub 2022 May 9. PMID 35534778